CLINICAL TRIAL: NCT06648018
Title: Fe-minine Health and Exercise
Brief Title: Comparison of Nutritional Information With Iron-succinate Supplementation in Healthy Women
Acronym: Fe-Health
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Primary Health Care Center, Region Östergötland (Unknown); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Fredrik H Nystrom, MD PhD full professor, senior consultant in internal medicine, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fe-minine health and exercise
Record Dates: First submitted 2024-09-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Well Being
Keywords: nutrition; exercise; iron; well being
MeSH Terms: conditions — Motor Activity | interventions — ferrous succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional information (Active Comparator): Written information about food with high iron content.
  Interventions: Behavioral: Nutritional information
- 100mg iron-succinate per day as a pill. (Experimental): Participants get 56 pills of 100mg iron-succinate to take one/day for 8 weeks.
  Interventions: Dietary Supplement: Iron-succinate

INTERVENTIONS:
Behavioral: Nutritional information — Written nutritional information about food with high content of iron.
  Arms: Nutritional information
Dietary Supplement: Iron-succinate — 100 mg of Iron-succinate per day.
  Arms: 100mg iron-succinate per day as a pill.

SUMMARY:
The primary aim of the current study is to evaluate the effects of dietary nutritional advice with regards to iron rich food sources or a daily oral supplement of 100 mg ferrous iron succinate in 80 menstruating, healthy women aged 20-40 years for 8 weeks. The study will use a randomized controlled non-blinded design, and 80 healthy women aged 20-40 years whom regularly exercise will be included. Data collection will be made through online, standardized forms using the digital platform REDCap 13.1.28 (Vanderbilt University, Nashville, TN, USA). Study personnel will register laboratory and body weight results through the same system. Participants will be randomized 1:1 to either follow written dietary recommendations to increase their dietary iron intake, or to use a daily oral supplement of 100 mg of iron succinate. Study parameters are blood tests (fasting blood samples will be collected by a licensed laboratory: serum iron, serum transferrin, serum transferrin saturation, serum ferritin, and serum soluble transferrin receptor, blood status (hemoglobin, MCV, MCH, MCHC, thrombocytes, leukocytes), and plasma high-sensitivity C-reactive protein (hsCRP) and Body height and weight as well as questionnaires.

DETAILED DESCRIPTION:
Aim The primary aim of the current study is to evaluate the effects of dietary nutritional advice with regards to iron rich food sources or a daily oral supplement of 100 mg ferrous iron succinate in 80 menstruating, healthy women aged 20-40 years.

Methods The study will use a randomized controlled non-blinded design, and 80 healthy women aged 20-40 years whom regularly exercise will be included. Data collection will be made through online, standardized forms using the digital platform REDCap 13.1.28 (Vanderbilt University, Nashville, TN, USA). Study personnel will register laboratory and body weight results through the same system.

Recruitment and participation criteria Individuals will be recruited through any or all of the following: at primary care center(s) in Sweden, via posters at the care center(s), via care providers during visits to the care center(s) and/or via external advertisement through social media and/or at public spaces.

Inclusion criteria will be menstruating women aged 20 to 40 years who are healthy and regularly exercise. As reimbursement, participants will receive 2000 SEK for the drawing of blood samples at the end of their study participation.

Inclusion visit

Individuals interested to participate will be booked for an inclusion visit with a study nurse during which oral and written information of the study will be provided, and a written consent will be given. Online, participants will then be asked to fill in the following information:

* A detailed online questionnaire regarding age, use of nicotine and tobacco products, and any drugs or supplements.
* A questionnaire on menstruation quantities including the number of menstruation days, the number of heavy menstruation days, and the menstrual product use, which has been shown to accurately estimate menstrual blood loss.24
* The Alcohol use disorders identification test (AUDIT)
* A food frequency questionnaire (FFQ)
* To evaluate physical activity, we will use the validated questions from the Swedish National Board of Health and Welfare,25 as well as the validated SED-GIH question of The Swedish School of Sport and Health Sciences (GIH) on sedentary behavior which was also developed with support from the Swedish National Board of Health and Welfare.26
* A questionnaire on gastrointestinal symptoms, including the number of bowel movements per week and the quality of them assessed using the Bristol stool scale (BSS). Gastrointestinal transit time can be approximated as defecation frequency, or more accurately, as stool consistency 27, and the BSS is one such questionnaire.

Body height and weight, with participants in light clothing without shoes, as well as fasting blood samples will be collected by a licensed laboratory: serum iron, serum transferrin, serum transferrin saturation, serum ferritin, and serum soluble transferrin receptor, blood status (hemoglobin, MCV, MCH, MCHC, thrombocytes, leukocytes), and plasma high-sensitivity C-reactive protein (hsCRP).

Intervention/control period Participants will be randomized 1:1 to either follow written dietary recommendations to increase their dietary iron intake, or to use a daily oral supplement of 100 mg of iron succinate.

Conclusion visit Of the above information, the following will be repeated after the conclusion of the 8 week intervention/control period: questionnaires on physical activity and gastrointestinal symptoms, the FFQ, and the drawing of blood samples.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria will be menstruating women aged 20 to 40 years who are healthy and regularly exercise.

-

Exclusion Criteria: Significant disease affecting inflammation and/or hemoglobin levels. Inability to cooperate or to fill out questionnaires.

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who are menstruating. This is a trial of potentially low ferritin levels in menstruating women.
Enrollment: 80 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Ferritin blood test | From enrollment to end of test period, 8 weeks.
  Change (increase) in serum ferritin levels.

SECONDARY OUTCOMES:
Changes in measures of hemoglobin | From enrollment to end of test period, 8 weeks.
  Changes in measures of hemoglobin levels by blood tests
Sense of well being and subjective sense of health | From enrollment to end of test period, 8 weeks.
  Sense of well being and subjective sense of health by questionnaires at start and baseline

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nyström, MD PhD Professor, Principal Investigator — Linkoeping University
Locations (1):
- Faculty of Medicine and Health Sciences Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
For ethical reasons such data will not be shared.